CLINICAL TRIAL: NCT00561093
Title: Pilot/Feasibility Randomized Control Trial to Examine the Effect of Oral Nutritional Supplements With Anti-inflammatory/Anti-oxidative Properties and Pentoxiphylline on Malnutrition-inflammation-cachexia Syndrome in Maintenance Hemodialysis Patients
Brief Title: Anit-Inflammatory and Anti-Oxidative Nutrition in Dialysis Patients
Acronym: AIONID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: DaVita, Inc. (Industry); Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21 DK78012 (completed); Harbor-UCLA LABioMed # 12630; R21DK078012 (NIH)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Hypoalbuminemia; Protein-energy Malnutrition; Inflammation; Oxidative Stress; Chronic Kidney Disease (CKD) Hemodialysis
Keywords: Hypoalbuminemia; Protein-energy malnutrition; Inflammation; Oxidative stress; Chronic Kidney disease (CKD) stage 5; maintenance hemodialysis
MeSH Terms: conditions — Hypoalbuminemia; Protein-Energy Malnutrition; Inflammation; Renal Insufficiency, Chronic | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Group A (n=25) Nepro (8 ounces) and Oxepa-similar anti-inflammatory module (2 ounces) AND pentoxiphylline (400 mg) while undergoing hemodialysis and the following non-dialysis day (6 days per week)
  Interventions: Drug: pentoxiphylline; Dietary Supplement: Nepro; Dietary Supplement: anti-inflammatory module (similar to Oxepa)
- B (Experimental): Group B (n=25) Nepro (8 ounces) and Oxepa-similar anti-inflammatory module (2 ounces) AND Placebo to imitate pentoxiphylline while undergoing hemodialysis and the following non-dialysis day (6 days per week)
  Interventions: Dietary Supplement: Nepro; Dietary Supplement: anti-inflammatory module (similar to Oxepa); Drug: Placebo pill imitating pentoxiphylline
- C (Experimental): Group C (n=25) Placebo dietary supplement to imitate Nepro (8 ounces) and Oxepa-similar anti-inflammatory module (2 ounces) AND pentoxiphylline (400 mg) while undergoing hemodialysis and the following non-dialysis day (6 days per week)
  Interventions: Drug: pentoxiphylline; Dietary Supplement: Placebo to imitate Nepro; Dietary Supplement: Placebo to imitate anti-inflammatory module (similar to Oxepa)
- D (Placebo Comparator): Group D (n=25) Placebo to imitate Nepro (8 ounces) and Oxepa-similar anti-inflammatory module (2 ounces) AND Placebo to imitate pentoxiphylline (400 mg) while undergoing hemodialysis and the following non-dialysis day (6 days per week)
  Interventions: Drug: Placebo pill imitating pentoxiphylline; Dietary Supplement: Placebo to imitate Nepro; Dietary Supplement: Placebo to imitate anti-inflammatory module (similar to Oxepa)

INTERVENTIONS:
Drug: pentoxiphylline — pentoxiphylline 400 mg daily, anti-inflammatory and appetite-stimulating while subjects undergo thrice weekly hemodialysis and during the following non-dialysis day (6 days per week)
  Other Names: Trental, 400 mg pills
  Arms: A; C
Dietary Supplement: Nepro — Nepro (8 ounces) one can while undergoing thrice weekly hemodialysis and during the following non-dialysis day (6 days per week)
  Other Names: Nepro with Carb ™ Steady
  Arms: A; B
Dietary Supplement: anti-inflammatory module (similar to Oxepa) — Oxepa-similar anti-inflammatory module (2 ounces) while undergoing thrice weekly hemodialysis and during the following non-dialysis day (6 days per week)
  Other Names: Oxepa-similar anti-inflammatory module (2 ounces)
  Arms: A; B
Drug: Placebo pill imitating pentoxiphylline — Placebo pill imitating pentoxiphylline 400 mg daily, to imitate the anti-inflammatory and appetite-stimulating pill while subjects undergo thrice weekly hemodialysis and during the following non-dialysis day (6 days per week)
  Other Names: Placebo pill imitating pentoxiphylline 400 mg daily, to imitate the anti-; inflammatory and appetite-stimulating pill while subjects undergo thrice; weekly hemodialysis and during the following non-dialysis day (6 days per week)
  Arms: B; D
Dietary Supplement: Placebo to imitate Nepro — Placebo to imitate Nepro (8 ounces), with less protein and calorie, one can while undergoing thrice weekly hemodialysis and during the following non-dialysis day (6 days per week)
  Other Names: Placebo to imitate Nepro (8 ounces), with less protein and calorie,
  Arms: C; D
Dietary Supplement: Placebo to imitate anti-inflammatory module (similar to Oxepa) — Placebo to imitate Oxepa-similar anti-inflammatory module (2 ounces), without anti-inflammatory or anti-oxidative ingredients, while undergoing thrice weekly hemodialysis and during the following non-dialysis day (6 days per week)
  Other Names: Placebo to immitate Oxepa-similar anti-inflammatory module (2 ounces), without anti-inflammatory or anti-oxidative ingredients,; 0011084880
  Arms: C; D

SUMMARY:
Study of efficiency and safety of oral nutritional supplements with anti-inflammatory and antioxidative properties combined with an appetite stimulant with anti-inflammatory properties (pentoxiphylline) in treatment of malnutrition-inflammation-cachexia syndrome in maintenance hemodialysis patients

DETAILED DESCRIPTION:
There are 350,000 hemodialysis patients in the USA; these are people who have end-stage kiney disease and whose survival depends on thrice weekly hemodialysis treatment in a dialysis clinic. Hemodialysis patients have an unacceptably high death rate, so that one out of every 4 to 5 patients die each year. Almost half of all deaths are believed to be from heart disease. Because markers of malnutrition and inflammation such as low amount of blood protein (serum albumin <4.0 g/dL), rather than traditional risk factors, are among the strongest predictors of early death and because malnutrition-inflammation appears to be closely related to oxidative stress in hemodialysis patients, we would like to examine that hypotesis that treating malnutrition-inflammation-oxidation by mean of nutritional support may improve outcomes in them. Low serum albumin <4.0 g/dL is observed in almost half of all hemodialysis patients and appears associated with low appetite, wasting, inflammation, malfunction of the vessels, cardiovascular disease and several fold increase in mortality.

We hypothesize that the malnutrition-inflammation can be significantly corrected by a simple in-center oral nutritional support with anti-inflammatory and antioxidant properties combined with an appetite stimulant with anti-inflammatory properties, leading to improved clinical and nutritional outcome measures in hemodialysis patients. We have proposed to the National Institutes of Health a pilot/feasibility study where dialysis patients will have 50-50 chance of receiving real treatment or a fake version of it (placebo). This method is called randomization, and this study type is called "randomized placebo-controlled clinical trial" with two arms, a so-called 2x2 factorial design. Our proposed study has a low-priced but efficient operational system and will be performed in 8 to 10 DaVita dialysis clinics in Los Angles area. During this 2-year pilot/feasibility study, we will test whether our proposed nutritional and anti-inflammatory treatments are safe and can improve low serum albumin and other relevant outcomes in 100 hemodialysis patients. Subjects will be adult hemodialysis patients with a serum albumin <4.0 g/dL.

The nutritional support arm will include a combination of 2 oral nutritional supplements; i.e., Nepro™ (8 oz), tailored for malnourished hemodialysis patients; and a condensed anti-inflammatory module similar to Oxepa™ (2 oz), designed for sick patients with inflammation and oxidative stress; or their placebos. The appetite stimulating arm will include a medication known as "pentoxifylline" (also known as Trental™) and the dose will be 400 mg daily or its placebo.

If a patient qualifies and agrees to participate in the study, there will be one month of observations and tests, followed by 16 weeks of treatment, and then one additional month of observation at the end. Both interventions are administered thrice weekly during routine hemodialysis for 16 weeks. Nutritional, inflammatory and oxidative measures, vessel wall (endothelial) function, quality of life and other clinical measures will be obtained before, during, and after the intervention. The safety and tolerability of the treatments, the feasibility of the study design, and the measurability of the outcomes will be examined.

We hope that the successful completion of this pilot/feasibility study in our campus leads to design of a large-scale clinical trial at the national level to improve survival in dialysis patients using nutritional and anti-inflammatory treatments.

Figure 1. Proposed pilot/feasibility study (see Appendix 1 for color version)

Group A (n=25) Nepro/Oxepa (2 cans) + PTX (400 mg) while on HD & the following day

Group B (n=25) Nepro/Oxepa (2 CANS) + placebo PTX while on HD& the following day

Group C (n=25) Placebo 2 cans + PTX (400 mg) while on HD& the following day

Group D (n=25) Placebo 2 cans + placebo PTX while on HD& the following day

PTX: pentoxifylline HD: Hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months on maintenance hemodialysis,
* Last 3-month averaged serum albumin <4.0 g/dl,
* Average monthly Kt/V>1.2,
* Dialysis time between 3 and 5 hours,
* Functioning AV graft or fistula or tunnel catheter that will not switch for 6 months,
* Standardized dialysis treatment per DaVita protocol.
* In case the averaged 3-month is not <4.0 g/dl but last month serum albumin <4.0 g/dl (worsening hypoalbuminemia) patient will be qualified, if 3-month averaged nPNA < 0.8 g/kg/day or a BMI < 20 kg/m2.

Exclusion Criteria:

* Peritoneal dialysis
* Terminal illnesses with life expectancy<6 months
* Maintenance hemodialysis less than 5 months
* Concurrent appetite stimulants
* Use of IDPN in the past 2-3 months
* Inability to follow and to comply with the instructions and guidelines
* Likelihood of pregnancy or intention to become pregnant
* Acute wasting condition or active systemic disease
* Pulse chemo therapy
* Non-compliance with dialysis treatment
* Dialysis catheter that may switch soon.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in serum albumin | 16 weeks

SECONDARY OUTCOMES:
Changes in body composition and measures of nutrition, inflammation, anemia, Health related quality of life (HRQOL), and tolerance | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kamyar Kalantar-Zadeh, MD MPH PhD, Principal Investigator — LABioMed at Harbor-UCLA; Arezu Dezfuli, MD, Study Director — LABioMed at Harbor-UCLA; Jennie Jing, MS, Study Director — LABioMed at Harbor-UCLA
Locations (2):
- United States (2):
  - DaVita Nutrition Services, Irvine, California
  - Los Angeles Biomedical Research Institute (LABioMed) at Harbor-UCLA, Torrance, California

REFERENCES:
- [Background] Kalantar-Zadeh K, Braglia A, Chow J, Kwon O, Kuwae N, Colman S, Cockram DB, Kopple JD. An anti-inflammatory and antioxidant nutritional supplement for hypoalbuminemic hemodialysis patients: a pilot/feasibility study. J Ren Nutr. 2005 Jul;15(3):318-31. doi: 10.1016/j.jrn.2005.04.004. PMID 16007562
- [Background] Colman S, Bross R, Benner D, Chow J, Braglia A, Arzaghi J, Dennis J, Martinez L, Baldo DB, Agarwal V, Trundnowski T, Zitterkoph J, Martinez B, Khawar OS, Kalantar-Zadeh K. The Nutritional and Inflammatory Evaluation in Dialysis patients (NIED) study: overview of the NIED study and the role of dietitians. J Ren Nutr. 2005 Apr;15(2):231-43. doi: 10.1053/j.jrn.2005.01.003. PMID 15827897
- [Background] Cooper A, Mikhail A, Lethbridge MW, Kemeny DM, Macdougall IC. Pentoxifylline improves hemoglobin levels in patients with erythropoietin-resistant anemia in renal failure. J Am Soc Nephrol. 2004 Jul;15(7):1877-82. doi: 10.1097/01.asn.0000131523.17045.56. PMID 15213276
- [Background] Kalantar-Zadeh K, Kilpatrick RD, Kuwae N, McAllister CJ, Alcorn H Jr, Kopple JD, Greenland S. Revisiting mortality predictability of serum albumin in the dialysis population: time dependency, longitudinal changes and population-attributable fraction. Nephrol Dial Transplant. 2005 Sep;20(9):1880-8. doi: 10.1093/ndt/gfh941. Epub 2005 Jun 14. PMID 15956056
- [Background] Kalantar-Zadeh K, Block G, McAllister CJ, Humphreys MH, Kopple JD. Appetite and inflammation, nutrition, anemia, and clinical outcome in hemodialysis patients. Am J Clin Nutr. 2004 Aug;80(2):299-307. doi: 10.1093/ajcn/80.2.299. PMID 15277149
- [Background] Kalantar-Zadeh K, Ikizler TA, Block G, Avram MM, Kopple JD. Malnutrition-inflammation complex syndrome in dialysis patients: causes and consequences. Am J Kidney Dis. 2003 Nov;42(5):864-81. doi: 10.1016/j.ajkd.2003.07.016. PMID 14582032
- [Background] Rammohan M, Kalantar-Zadeh K, Liang A, Ghossein C. Megestrol acetate in a moderate dose for the treatment of malnutrition-inflammation complex in maintenance dialysis patients. J Ren Nutr. 2005 Jul;15(3):345-55. doi: 10.1016/j.jrn.2004.10.006. PMID 16007564
- [Background] Kalantar-Zadeh K, Balakrishnan VS. The kidney disease wasting: inflammation, oxidative stress, and diet-gene interaction. Hemodial Int. 2006 Oct;10(4):315-25. doi: 10.1111/j.1542-4758.2006.00124.x. PMID 17014506
- [Background] Kalantar-Zadeh K. Recent advances in understanding the malnutrition-inflammation-cachexia syndrome in chronic kidney disease patients: What is next? Semin Dial. 2005 Sep-Oct;18(5):365-9. doi: 10.1111/j.1525-139X.2005.00074.x. PMID 16191172
- [Background] Kalantar-Zadeh K, Stenvinkel P, Bross R, Khawar OS, Rammohan M, Colman S, Benner D. Kidney insufficiency and nutrient-based modulation of inflammation. Curr Opin Clin Nutr Metab Care. 2005 Jul;8(4):388-96. doi: 10.1097/01.mco.0000172578.56396.9e. PMID 15930963
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133